CLINICAL TRIAL: NCT04622241
Title: Impact of Housing Modifications Combined With Piperonyl Butoxide (PBO) Long-lasting Insecticidal Nets (LLINs) on the Malaria Burden in Uganda: a Cluster-randomised Trial
Brief Title: Uganda Housing Modification Study
Acronym: UHMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Infectious Diseases Research Collaboration, Uganda (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); United States Agency for International Development (USAID) (U.S. Federal Agency); London School of Hygiene and Tropical Medicine (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 72061720FA00002
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Malaria; Anemia
Keywords: Housing Modification; Vector Control; Uganda; Malaria Control
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Intervention Model Description: Phase II will be carried out as a cluster-randomized trial with 3 arms (2 interventions selected from the pilot study, and 1 control). There will be 20 clusters per arm (60 clusters total) and a cluster will be defined as an enumeration area within a village. All participating households in the selected clusters will have PBO LLINs, and households in intervention clusters will also receive the specified housing modifications. The impact of the interventions on malaria burden will be assessed through a cohort study, cross-sectional community surveys, entomology surveillance, a qualitative study, and an economic evaluation. The primary outcome of the trial will be clinical malaria incidence in children aged < 60 months.
Masking Description: Masking is not possible due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Eave Tubes - Traditional House (Experimental): Installation of eave tubes in traditional homes.
  Interventions: Other: Eave Tubes
- Eave Tubes - Modern House (Experimental): Installation of eave tubes in modern homes.
  Interventions: Other: Eave Tubes
- Eave Ribbons - Traditional House (Experimental): Installation of eave ribbons in traditional homes.
  Interventions: Other: Eave Ribbons
- Eave Ribbons - Modern House (Experimental): Installation of eave ribbons in modern homes.
  Interventions: Other: Eave Ribbons
- Full House Screening - Traditional House (Experimental): Installation of full house screening, includes screening eaves and windows, in traditional homes.
  Interventions: Other: Full House Screening
- Full House Screening - Modern House (Experimental): Installation of full house screening, includes screening eaves and windows, in modern homes.
  Interventions: Other: Full House Screening
- Partial House Screening - Traditional House (Experimental): Installation of partial screening, includee either screening of the eaves or installing a screened ceiling, in traditional homes.
  Interventions: Other: Partial House Screening
- Partial House Screening - Modern House (Experimental): Installation of partial screening, includee either screening of the eaves or installing a screened ceiling, in modern homes.
  Interventions: Other: Partial House Screening
- Control - Traditional House (No Intervention): Control group with no intervention in traditional homes
- Control - Modern House (No Intervention): Control group with no intervention in modern homes.

INTERVENTIONS:
Other: Eave Tubes — The eave tubes are PVC tubes with a diameter of 15 cm installed in the outer wall of occupied rooms (e.g. bedrooms and living rooms but not storage rooms) at 1.5-2 m intervals, fitted with electrostatic mesh inserts coated with insecticides. No additional screening will be done. All households will be provided with piperonyl butoxide (PBO) long-lasting insecticidal nets (LLINs) - one for every two residents.
  Arms: Eave Tubes - Modern House; Eave Tubes - Traditional House
Other: Eave Ribbons — Eave ribbons are 15 cm-wide triple-layered hessian fabrics (burlap-line fabric woven from sisal fibres, procured locally), in lengths starting 1 m that can be attached to houses using nails, adhesives or Velcro, without completely closing eave-spaces. The eave ribbons will be treated by study staff with a commonly used spatial repellent, transfluthrin. Eave ribbons will be retreated by study staff after 6 months (only in Phase II, if selected for inclusion in the cluster-randomised trial).
  All households will be provided with piperonyl butoxide (PBO) long-lasting insecticidal nets (LLINs) - one for every two residents.
  Arms: Eave Ribbons - Modern House; Eave Ribbons - Traditional House
Other: Full House Screening — Full house screening includes screening eaves/ceilings, ventilation openings, and windows. Eaves/ceiling, air vents, and windows of eligible houses will be screened with wire mesh or other locally available screening materials. or ceilings, if eaves are closed" and ventilation openings. We are also filling in any gaps in the walls. All households will be provided with piperonyl butoxide (PBO) long-lasting insecticidal nets (LLINs) - one for every two residents.
  Arms: Full House Screening - Modern House; Full House Screening - Traditional House
Other: Partial House Screening — Partial screening will include either screening of the eaves or installing a screened ceiling, where no ceiling is present. In traditional houses, a netting (either insecticide-impregnated or untreated) may be either fixed in multiple places in the rafters or by hanging from a single central point and attached to the walls. No other screening or filling of the gaps will be done in partially screened houses.All households will be provided with piperonyl butoxide (PBO) long-lasting insecticidal nets (LLINs) - one for every two residents.
  Arms: Partial House Screening - Modern House; Partial House Screening - Traditional House

SUMMARY:
To explore housing modification as a malaria control intervention, and to assess the degree to which it may offer protection in moderate to high malaria endemicity settings, we propose a two-phase study evaluating epidemiological and entomological effectiveness, cost-effectiveness, feasibility, and acceptability of housing modification in Uganda. The first phase will be a pilot implementation assessing the feasibility of candidate housing modification interventions, followed by a cluster randomised control trial of the most effective, scalable, and cost-effective interventions.

DETAILED DESCRIPTION:
The study will be conducted in two phases, beginning with a pilot (Phase I). The aim of the pilot will be to develop and test four types of housing modifications in both modern houses (those with brick or stone walls) and traditionally constructed houses (those with mud walls). The housing modifications will include: (1) full house screening (eaves and windows), (2) partial house screening (eaves or ceiling), (3) eave tubes, and (4) eave ribbons. Community input will be sought during the development of the housing prototypes.

In the pilot, all 4 interventions will be implemented in both modern and traditional houses, plus a control arm in each group. All households will have access to PBO LLINs. Community input will be sought during the development of the housing prototypes. The pilot will include 10 arms in total, each consisting of 20 households, equal to 200 households (160 in the intervention and 40 in the control arm) in total. The feasibility and effectiveness of the interventions will be assessed through a qualitative study (FGDs and interviews), evaluation of the costs and implementation of the interventions, and entomology surveys (using CDC light traps). One to two housing interventions will be selected for Phase II following the review and discussion of the pilot results with the trial steering committee.

Phase II will include a cluster-randomised trial. A cluster will be defined as a village (or segment of a village consisting of ~100 households). In the cluster-randomised trial, up to 2 interventions vs 1 control arm will be assessed in 20 clusters per arm (60 clusters total). The clusters will be non-contiguous, with a buffer zone of 300-500m. All households in the selected clusters will have PBO LLINs; households in intervention clusters will also receive the specified housing modifications. The impact of the interventions will be assessed through a cohort study, cross-sectional community surveys, entomology surveillance, a qualitative study, and an economic evaluation. The primary outcome of the trial will be clinical malaria incidence in children aged < 60 months as measured in the cohort study.

ELIGIBILITY:
Phase I

Inclusion criteria

* At least one adult aged 18 years or older present
* Agreement of the adult resident to provide informed consent for the pilot study

Phase II

Cohort Study

Inclusion Criteria:

* Household considered their primary residence
* Child aged less than 59 months
* Agreement to come to the study clinic for any febrile illness
* Agreement to avoid antimalarial medications outside the study
* Provision of written informed consent (for parent or guardian in case of children)

Cross-sectional Community Survey - Household Survey

Inclusion Criteria:

* At least one household resident between 6 months and 14 years of age present (with an adult caregiver willing to provide informed consent for the clinical survey)
* At least one adult aged 18 years or older present
* Adult is a usual resident who slept in the sampled household on the night before the survey
* Agreement of the adult resident to provide informed consent for the household survey

Exclusion Criteria:

* Dwelling destroyed or not found
* Household vacant
* No adult resident home on more than 3 occasions

Cross-sectional Community Survey - Clinical Survey

Inclusion Criteria:

* Child aged 6 months to 14 years
* Usual resident who was present in the sampled household on the night before the survey
* Agreement of parent/guardian to provide informed consent
* Agreement of child aged 8 years or older to provide assent

Exclusion Criterion:

* Child not home on day of survey

Recruitment of Field Workers for entomology activities (human landing catches).

Inclusion Criteria:

* Willingness to take chemoprophylaxis for malaria
* Willingness to abstain from alcohol during working hours
* No significant past medical history.

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2422 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of malaria | 12 months following housing modification
  Number of incident episodes of clinical malaria per time of observation. Incident episodes of malaria defined as any treatment for malaria > 14 days after any prior treatment for malaria

SECONDARY OUTCOMES:
Parasite prevalence | 12 months following housing modification
  Proportion of study participants with a thick blood smear positive for asexual parasites as measured by microscopy
Prevalence of anaemia | 12 months following housing modification
  Proportion of haemoglobin measurements categorised as anaemia as per WHO age-stratified guidelines
Vector density | 12 months following housing modification
  Number of female Anopheles mosquitoes captured/room per night by CDC light traps
Sporozoite rate | 12 months following housing modification
  Proportion of captured female Anopheles mosquitoes that test positive for sporozoites
Annual entomological inoculation rate | 12 months following housing modification
  Number of infected bites per person per year (human biting rate x sporozoite rate x 365 days/year)
Proportion of mosquitoes with insecticide resistance | 12 months following housing modification
  Proportion of mosquitoes with phenotypic expression of insecticide resistance or containing genetic polymorphisms associated with resistance to insecticides of interest as identified by PCR
Proportion of individuals satisfied with the interventions | 12 months following housing modification
  Indicator of acceptability
Proportion of households that require minimal maintenance of the implemented intervention over the period of the study, by study intervention | 12 months following housing modification
  Indicator of durability
Longer term cost of the maintenance and upkeep of the implemented intervention, by study intervention | 12 months following housing modification
  Indicator of durability
Costs of housing improvements, including maintenance, by improvement type | 12 months following housing modification
  Indicator of feasibility
Incremental cost-effectiveness ratios (ICER) of each package | 12 months following housing modification
  Cost per malaria case averted, Cost per DALY averted
Proportion of households that received the assigned housing modification | 12 months following housing modification
  Indicator of fidelity
Proportion of households that received 1 PBO LLIN for every 2 residents | 12 months following housing modification
  Indicator of fidelity
Proportion of households that received full/partial/no housing modifications | 12 months following housing modification
  Dose delivered
Proportion of households that received adequate/inadequate/no PBO LLINs | 12 months following housing modification
  Dose delivered
Proportion of households that utilized full/partial/no housing modifications | 12 months following housing modification
  Dose received
Proportion of household residents that slept under a PBO LLIN the previous night | 12 months following housing modification
  Dose received
Proportion of households that were fully covered by the assigned housing modification | 12 months following housing modification
  Indicator of reach
Proportion of household residents that were fully covered by the PBO LLINs | 12 months following housing modification
  Indicator of reach
  Proportion of households fully covered by both the modifications & PBO LLINs
Proportion of households fully covered by both the modifications & PBO LLINs | 12 months following housing modification
  Indicator of reach

CONTACTS AND LOCATIONS:
Overall Officials: Nelli Westercamp, PhD MBA, Principal Investigator — Centers for Disease Control and Prevention; Moses Kamya, MBChB PhD, Principal Investigator — Infectious Diseases Research Collaboration
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snyman K, Ochieng W, Gonahasa S, Aber J, Katureebe A, Staedke SG, Kamya MR, Westercamp N, Pitt C. Housing modification to prevent malaria in Uganda: an analysis of costs, willingness to pay, and equity. Malar J. 2025 Dec 24. doi: 10.1186/s12936-025-05757-0. Online ahead of print. PMID 41444546
- [Derived] Kayendeke M, Nabirye C, Nayiga S, Westercamp N, Gonahasa S, Katureebe A, Kamya MR, Staedke SG, Hutchinson E. House modifications as a malaria control tool: how does local context shape participants' experience and interpretation in Uganda? Malar J. 2023 Aug 25;22(1):244. doi: 10.1186/s12936-023-04669-1. PMID 37626312